CLINICAL TRIAL: NCT07278453
Title: Optimal Tuberculosis Screening and Tuberculosis Preventive Therapy Delivery Strategies to Improve Maternal and Birth Outcomes Among Pregnant Women With HIV in Uganda: a Randomized Trial
Brief Title: TB SCReening Improves Preventive Therapy Uptake in Pregnant Women With HIV
Acronym: TB SCRIPT-Moms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R61HL178398 (NIH); R61HL178398 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pregnant HIV Positive Women; HIV; Tuberculosis (TB)
Keywords: pregnant women with HIV; pregnant women; hiv; tuberculosis; screening; tuberculosis preventive therapy
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO 4-part symptom screening (TB screening control arm) (Other): In the TB screening trial, participants will be randomized to one of two WHO-recommended TB screening strategies: symptom-based TB screening (current practice) or CRP-based TB screening. Participants randomized to symptom-based screening will be screened by study staff using the WHO 4-part symptom screen (W4SS). Participants randomized to the W4SS arm who report ≥1 TB symptom (current cough, fever, night sweats, weight loss/inappropriate weight gain) in the past 30 days will be regarded as TB screen-positive. Participants randomized to the W4SS arm who none of the 4 TB symptoms in the past 30 days will be regarded as TB screen-negative.
  Interventions: Diagnostic Test: CRP screening (TB screening intervention arm)
- Immediate TPT (TPT control arm) (Other): In the TB preventive therapy (TPT) delivery trial, participants will be randomized to either immediate (antepartum) TPT (current recommendation) or deferred (postpartum) TPT, where TPT is deferred to 4 weeks postpartum. Participants randomized to immediate TPT will immediately initiate TPT (while pregnant), in accordance with current WHO TPT recommendations for pregnant women with HIV.
  Interventions: Other: Deferred TPT (TPT delivery trial intervention arm)

INTERVENTIONS:
Diagnostic Test: CRP screening (TB screening intervention arm) — In the TB screening trial, participants will be randomized to one of two WHO-recommended TB screening strategies: symptom-based TB screening (current practice) or CRP-based TB screening. Participants randomized to CRP-based screening will have CRP concentrations measured by study staff at the point-of-care, using blood obtained by finger prick. Participants randomized to the CRP arm with CRP ≥5 mg/L will be regarded as TB screen-positive. Participants randomized to the CRP arm with CRP <5 mg/L will be regarded as TB screen-negative.
  Arms: WHO 4-part symptom screening (TB screening control arm)
Other: Deferred TPT (TPT delivery trial intervention arm) — In the TB preventive therapy (TPT) delivery trial, participants will be randomized to either immediate (antepartum) TPT (current recommendation) or deferred (postpartum) TPT, where TPT is deferred to 4 weeks postpartum. Participants randomized to deferred TPT will initiate TPT 4 weeks after delivery.
  Arms: Immediate TPT (TPT control arm)

SUMMARY:
Because pregnant women have been excluded from clinical research, including tuberculosis (TB) research, little is known about diagnosing, treating and preventing TB in pregnant women. We plan to perform a two-stage randomized trial that will identify best practices for screening pregnant and postpartum women for active TB (screening by symptoms vs. C-reactive protein levels) and the optimal timing of TPT initiation, relative to pregnancy (immediately during pregnancy or deferred to postpartum). Because undiagnosed TB among pregnant women with HIV is associated with many devastating complications to both the mother and fetus, this research has the potential to improve maternal and birth outcomes worldwide.

ELIGIBILITY:
For the TB screening trial, eligible patients include pregnant women with a viable singleton pregnancy by ultrasound, confirmed HIV infection, no current or planned TB treatment, no treatment with a drug with anti-mycobacterial activity within the past 2 weeks, no history of TB treatment or TPT within the past 2 years, lives within 20 km of the enrollment site, plans to deliver at the enrollment site, no plans to transfer antenatal care to a non-participating clinic, and no signs or symptoms of early or active labor.

For the TPT delivery trial, eligible participants are participants in the TB screening trial who screened negative for TB by their randomization assignment, are eligible for TPT, are not taking any drug contraindicated for use with rifamycins, are not a contact with a TB case with known drug resistance to isoniazid or rifampin, are not heavy or binge alcohol consumers, do not have a history of liver disease, do not have liver enzymes ≥3-times the upper limit of normal.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of TB cases detected | Up to 6 months postpartum
  The primary outcome for the TB screening trial is the proportion of TB cases detected by baseline and repeated rounds of TB screening, up to 6-months postpartum
Composite safety outcome | Up to 28 days postpartum
  The primary safety outcome of the TPT delivery trial is the composite endpoint that includes spontaneous abortion, stillbirth, low birthweight, preterm birth and neonatal death
Composite effectiveness outcome | Up to 2-years after TPT initiation
  The primary effectiveness outcome of the TPT delivery trial is a composite endpoint of maternal 2-year TB incidence and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Yoon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kampala Capital City Authority (KCCA) clinics, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No